CLINICAL TRIAL: NCT06799767
Title: Implementation Of Radiological Diagnostics In Patients With Deep Endometriosis
Brief Title: Radiological Diagnostics in Patients With Deep Endometriosis
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Endo-RAD
Record Dates: First submitted 2024-11-28; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-11

CONDITIONS: Deep Endometriosis
Keywords: deep endometriosis; radiological diagnostics; tractography; augmented reality; 3D-modelling; radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Endometriosis is a benign, chronic, recurrent disease characterised by the presence of endometrial glands and stroma outside the uterine cavity. A non-negligible proportion of patients, 2-37%, are affected by deep endometriosis (DIE), defined as the pathology's involvement of the muscular tunic propria of the abdomino-pelvic organs.

From a therapeutic point of view, a medical or surgical approach is possible. The choice is influenced by several factors, such as the patient's age, reproductive desire, the extent of symptoms, the size and location of the endometriosis lesions, and the presence of organ damage. Although the surgical approach brings satisfactory results in terms of symptom reduction and improved fertility, the risk of complications can be very high, especially in the case of DIE, as bladder, rectal and sexual function can be compromised due to iatrogenic damage to the autonomic fibres that innervate the pelvic organs. Recently, the concept of 'nerve-sparing' surgery has been extended to gynaecology, and in particular to surgery for the treatment of endometriosis, showing encouraging results in terms of both symptom control and functional outcome.

In recent years, nuclear magnetic resonance imaging (NMR) has been increasingly helpful in the diagnosis of endometriosis and adenomyosis and is increasingly used in pre-operative planning.

DETAILED DESCRIPTION:
Endometriosis is a benign, chronic, recurrent condition characterised by the presence of endometrial glands and stroma outside the uterine cavity. Although most frequently localised at the ovarian level (17 - 44%), a proportion of 2-37% of patients are affected by deep endometriosis (DIE), which involves the muscular tunic propria of the abdomino-pelvic organs. The most commonly affected sites are the rectovaginal septum, utero-sacral ligaments, rectum and sigma, ureters, parameters, hypogastric nerves, bladder and pre-vesical peritoneum.

In recent years, nuclear magnetic resonance imaging (NMR) has been increasingly helpful in the diagnosis of endometriosis and adenomyosis and is increasingly used in pre-operative planning together with transvaginal and/or transabdominal ultrasound. Recently, new techniques have been developed, such as Diffusion Tensor Imaging (DTI), Diffusion Weighted Imaging (DWI) and Dynamic Contrast Enhanced (DCE), whose gynaecological applications are currently in their infancy.

The study aims to evaluate the diagnostic accuracy and applicability of new MRI techniques in patients with deep endometriosis and candidates for surgical treatment.

In particular, the techniques that the investigators intend to investigate are: augmented reality, tractography, 3D-modelling, radiomics.

The use of these innovative methods, based on MRI techniques, may make it possible not only to plan an even more personalised treatment approach, selecting patients who could benefit from different treatments (such as presacral neurectomy, nerve root infiltration neurostimulation and the use of effective analgesics for neuropathic pain), but also to facilitate the localisation of endometriotic lesions during laparoscopic surgery, allowing the surgeon to assess their relationship with the main nerve and vascular structures of the pelvis and increasingly facilitating the nerve-sparing approach.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and ultrasound diagnosis of deep endometriosis, with or without ovarian endometriosis, with indication for MRI for further diagnosis and subsequent candidate for laparoscopic surgical treatment of the pathology
* Age between 18 and 40 years
* Obtaining informed consent

Exclusion Criteria:

* Previous abdominal surgery
* Personal history of malignancy (current or previous)
* Chronic inflammatory bowel disease (Crohn's disease, Ulcerative Rectocolitis, Indeterminate Colitis), interstitial cystitis
* Personal history of Pelvic Inflammatory Disease (PID), active or previous
* Previous radiotherapy/chemotherapy
* Radiculopathy, herniated discs, spinal abnormalities and pathologies
* Laparotomic conversion during surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a clinical and ultrasound diagnosis of deep endometriosis who are candidates for MRI for further diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostics and the applicability of new MRI techniques: tractography | During the first visit after enrollment
  Assessing sacral plexus root abnormalities by DTI-RMN and analysing the correlation between DTI abnormalities and the presence and severity of typical endometriosis symptoms (chronic pelvic pain, dysmenorrhoea, dyspareunia, ovulatory pain, dyschezia and dysuria) through Numerical Rating Scale (NRS), that is 0 "no pain," 10 "worst pain imaginable".
Diagnostic accuracy and applicability of new MRI techniques: augmented reality | During the first visit after enrollment
  Evaluate the diagnostic accuracy and precision of fiber tractography (FT) in reconstructing the course of the ureters bilaterally and mapping the hypogastric nerve bilaterally by comparing images obtained on MRI with in vivo surgical dissection
Diagnostic accuracy and applicability of new MRI techniques: 3D-modelling | During the first visit after enrollment
  Evaluate the diagnostic accuracy of 3D models of endometriosis nodules of the rectum and sigma obtained by MRI
Diagnostic accuracy and applicability of new MRI techniques: radiomics | During the first visit after enrollment
  Develop a pattern-recognition system based on MRI techniques for the histological nature (stromal vs. fibrotic) of the endometriosis nodules examined. Confirmation will be obtained on the basis of the definitive histological examination after surgery

SECONDARY OUTCOMES:
Diagnostics and the applicability of new MRI techniques: tractography | During surgery
  Assessing the correlation between DTI abnormalities and the location of endometriotic lesions found during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Renato Seracchioli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy